CLINICAL TRIAL: NCT03042390
Title: Multicenter Retrospective Study of the Effectiveness and Safety of Darunavir/Cobicistat (DRV/c) Containing Regimens in Routine Clinical Practice
Brief Title: Study of the Effectiveness and Safety of Darunavir/Cobicistat (DRV/c) Containing Regimens in Routine Clinical Practice
Acronym: CoDAR
Status: Completed | Type: Observational
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: GESIDA 9316
Record Dates: First submitted 2016-12-19; First posted 2017-02-03 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2016-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DArunavir/cobicistat: Patients starting treatment with a regimen containing Darunavir / cobicistat for at least 24 weeks

SUMMARY:
This is a retrospective observational study of patients who have taken a regimen containing DRV / c at least 24 weeks prior to study initiation

DETAILED DESCRIPTION:
The study will include 750 patients and will record data at 24 weeks. The study will also record data at 48 weeks for those patients whom these data are available

ELIGIBILITY:
Inclusion Criteria:

* Patients with HIV infection
* Inform consent document.
* To have initiated therapy containing DRV / c and have a follow-up of at least 24 Weeks.

Exclusion Criteria:

* Not having evaluable clinical data of the patient
* Patients not routinely followed in the center
* Patient less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients that initiated treatment with a régimen containing DRV/c at least 24 weeks prior initiation of study.
Sampling Method: Non-Probability Sample
Enrollment: 762 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Virological effectiveness data: Percentage of patients with undetectable viral load | 24 weeks
  Virological effectiveness data at 24 weeks: Percentage of patients with undetectable viral load, defined as HIV RNA <50 copies / m.
Virological effectiveness data: change in the number of CD4 + T cells at 24 weeks | 24 weeks
  Change in the number of CD4 + T cells at 24 weeks
Virological effectiveness data: time to loss of virological efficacy. | 24 weeks
  Defined virological failure as two consecutive levels of HIV RNA > 50 copies / mL or single HIV RNA ≥ 500 copies / mL

SECONDARY OUTCOMES:
Virological effectiveness data: Percentage of patients with undetectable viral load, defined as HIV RNA levels ≤ 50 copies / mL or limit of detection of the center, at 48 weeks | 48 weeks
  Virological effectiveness data at 48 weeks
Virological effectiveness data: change in the number of CD4 + T cells, at 48 weeks | 48 weeks
  Virological effectiveness data at 48 weeks: change in the number of CD4 + T cells
Changes in the renal profile: Comparison of mean values of Creatinine and eFG (CKD-EPI). | Basal and 24 weeks/48 weeks
  Creatinine (mg/dl), eFG (CKD-EPI) (ml/min/1,73 m2),
Changes in the lipid profile: Comparison of mean values of total cholesterol values, Col LDL, Col HDL and TG. | basal and 24 weeks/48 weeks
  Units: mg/dl or mmol/l
Changes in the hepatic profile: comparison of mean values of GOT, GPT, FA, GGT and BrT | basal and 24 weeks/48 weeks
  GOT, GPT, FA, GGT in units: UI/l or μKat/l or mU/ml. BrT in units: mg/dl or micromol/l
Tolerability data:Rate of patients discontinuing treatment for toxicity. | 24 weeks/48 weeks
  Toxicity to the treatment or virological failure
Tolerability data: Rate of patients discontinuing treatment for virological failure at 24 weeks / 48 weeks | 24 weeks/48 weeks
  Virological failure defined as two consecutive levels of HIV RNA > 50 copies / mL or single HIV RNA ≥ 500 copies / mL
Rate of patients who develop any adverse effects:frequency of adverse events,frequency of serious adverse events, frequency of adverse events leading to discontinuation of treatment, number of deaths and frequency of laboratory abnormalities. | 24 weeks/48 weeks
Representative subgroups of patients according to the treatment that patient is taking: Percentage of patients with different Darunavir/cobicistat based regimens (Monotherapy, Bitherapy, triple Therapy, others) | 24 weeks / 48 weeks
Provenance treatments: Percentage of patients with different prior therapies (Darunavir Therapy, Other PI therapies, NNRTI based regimen, INI bases regimen | 24 weeks / 48 weeks
Reason for the change prior the initiation:Percentage of patients with each main reason to change to a DRV/c based regimen (first regimen, simplification, intolerance or toxicity, prior adherence problems, prior interactions, prior failure, others) | 24 weeks / 48 weeks

CONTACTS AND LOCATIONS:
Locations (20):
- Spain (20):
  - Hospital Costa del Sol, Málaga, Marbella
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital del Vall d'Hebron, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital de Guadalajara, Guadalajara
  - Hospital Infanta Leonor, Madrid
  - Hospital La Paz, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Príncipe de Asturias, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital de Son Llatzer, Palma de Mallorca
  - Hospital de Valme, Seville
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital Clínico de Valencia, Valencia
  - Hospital La Fe, Valencia
  - Complejo Hospitalaria Alvaron Cunqueiro, Vigo

REFERENCES:
- [Derived] Perez Elias MJ, Alejos B, Gutierrez MM, Crespo M, De Los Santos Gil I, Ribera E, Galindo MJ, Lozano F, Payeras Cifre A, Boix V, Montero-Alonso M, Sanz J, De La Torre Lima J, Palacios R, De La Fuente Moral S, Martinez E; Codar Study Group. Dynamics of creatinine estimated glomerular filtration rate using one or more antiretrovirals that inhibit creatinine tubular secretion. J Antimicrob Chemother. 2021 Mar 12;76(4):1046-1050. doi: 10.1093/jac/dkaa547. PMID 33501995
- [Derived] Perez Elias MJ, Alejos B, Vivancos MJ, Ribera E, Galindo MJ, Vilanova-Trillo L, Garcia-Fraile Fraile LJ, de La Fuente Moral S, Garcia De Lomas J, Lozano F, Mateo Garcia MG, Tasias Pitarch M, Diez Martinez M, Rojas J, Raya-Cruz M, Sepulveda MA, Troya J, Del Campo S, Martinez E; CODAR study group. Outcomes by sex following treatment initiation with darunavir/cobicistat in a large Spanish cohort of the CODAR study (GeSIDA 9316). J Antimicrob Chemother. 2019 Oct 1;74(10):3044-3048. doi: 10.1093/jac/dkz254. PMID 31236601